CLINICAL TRIAL: NCT01619215
Title: The Effects of Bariatric Surgeries on Non-Alcoholic Fatty Liver Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: King Saud University (Other)
Responsible Party: Principal Investigator, Mazen Hassanain, Assistant Professor & consultant HPB and Transplant surgeon, King Saud University
Other Study IDs: KSULDRCBSMH001
Record Dates: First submitted 2012-05-27; First posted 2012-06-14 (Estimated); Last update posted 2018-03-30 (Actual); Status verified 2018-03

CONDITIONS: Obesity, Morbid; Non-Alcoholic Fatty Liver Disease
MeSH Terms: conditions — Obesity, Morbid; Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood (serum, plasma, and RNA isolate) Liver core biopsy Subcutaneous fat Visceral fat Abdominal wall muscle
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Bariatric Surgery: As the number of patients dropping out during follow-up, we had difficulty achieving our secondary outcomes, and so the team decided to continue the recruitment until all our outcomes are reached. Main part of the primary outcomes is finalised and published The effects of bariatric surgeries on nonalcoholic fatty liver disease. Aldoheyan T, Hassanain M, Al-Mulhim A, Al-Sabhan A, Al-Amro S, Bamehriz F, Al-Khalidi H. Surg Endosc. 2016 Jul 12

SUMMARY:
Non-alcoholic fatty liver disease (NAFLD) is the most common form of chronic liver disease. In the absence of chronic alcohol abuse or other liver diseases, NAFLD incorporates a wide spectrum of liver pathologies and is defined by fatty infiltration of the liver (simple hepatosteatosis). It can progress to non-alcoholic steatohepatitis (NASH) and later fibrosis, cirrhosis, and eventually some patients may develop hepatocellular carcinoma with or without cirrhosis. The exact cause of NAFLD is yet to be cleared and it is, therefore, an active area for research. The diagnosis of NAFLD is achieved through histological examination of liver biopsies (invasive), non-invasive markers using serum biomarkers and imaging techniques are still under development. Pathological diagnosis can be then subcategorized based on several scoring systems. More widely used are the Brunt Score or NAS (NAFLD activity score) and the Kleiner's modified NAS.

Obesity is highly associated with NAFLD, as the epidemic of obesity has made NAFLD more prevalent. In addition insulin resistance has been linked to NAFLD and this is explained by the increased influx of free fatty acids (FFAs) into the liver. FFA undergoes either β-oxidation or esterification with glycerol to form triglycerides (TGs), resulting in an additional source of fat in the liver. Due to the strong association of NAFLD with obesity, weight reduction procedures are used for the management of NAFLD. In fact, this has been shown to be effective by several studies. However, other studies have reported liver deterioration after bariatric intervention. This conflict is what makes the effects of bariatric procedures a challenging field for further studies. Consequently in this study we are aimed to examine histologic, metabolic and liver function changes induced by the different therapeutic bariatric procedures.

DETAILED DESCRIPTION:
35 consecutive patients referred for bariatric surgery will be recruited either at the obesity clinic, or from inpatient (scheduled for bariatric surgery). A detailed history and a complete physical examination will be done at the first visit along with anthropometric measures; routine blood tests, liver function, hormonal assessment, and certain metabolic and inflammatory markers will be evaluated. They will also have an abdominal ultrasound for initial NAFLD assessment, fibroscan to detect liver fibrosis, and an MRI to measure hepatic fat content and body fat composition including intra-abdominal and extra-abdominal fat. These patients will be asked to lose a certain amount of kilos (depending on their BMI and the surgeon preference) out of their original weight, in order to become candidates for bariatric surgery at King Saud University Hospital (KKUH).

At the second visit, (if they lose the recommended amount weight) we will assess their weight loss; obtain blood for the same hormonal and inflammatory markers assessment. Nonetheless, if they did not lose weight and the treating surgeon gave them a third appointment, we will consider their third visit as a second visit; preforming all the investigations mentioned above. In this case we will interpret their results with respect to the total duration of "before surgery" weight loss.

During the operation, tissue biopsy will be taken with a core needle biopsy for the liver and a sharp non-thermal instrument for subcutaneous fat, visceral fat, and abdominal muscle immediately after skin incision. A CAP certified tissue manager would process all tissues. Liver biopsy will be sliced it to two parts; the first half is for histological evaluation, but the other half will be stored for tissue studies. The histologic slides will be stained with hematoxylin and eosin (H&E), and Masson Trichrome stains for microscopic evaluation. This evaluation will be provided by a single histopathologist who will be blinded to the patients' clinical condition, and the order of the biopsy.

Follow Up:

After the surgery follow up appointments will be scheduled 3 months, 6 months, 1 year, and annually till 5 years. The followings will be done in each visit:

1. Thorough physical exam as per the CRF.
2. Take a blood sample to evaluate liver function, metabolic, and inflammatory changes using the same parameters as those in the baseline.
3. Request for: fibroscan and abdominal ultrasound. Second, third and fourth liver biopsies will be taken percutaneously 3 months, 1 year, and 5 years following the initial biopsy respectively. These biopsies will be obtained using core tissue biopsy with ultrasound guidance for the same histological assessment and tissue studies. Another MRI will be schedule 1 year after the surgery.

Specimens collected under this trial will be part of the King Saud University Liver Disease Research Centre Biobanking and will follow all policy and procedures within the biobanking protocol as approved by the IRB committee.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 to 60 years.
* Eligible for obesity surgery according to the following criteria:

  * BMI > 30 kg/m2.
  * Ability to demonstrate eating habit control by reducing 10% of the original weight prior to surgery
  * Pass the nutritional and the psychological assessment
  * Pass the preoperative testing to determine the operative risk
* Ultrasound diagnosis of NAFLD prior to surgery.
* Written informed consent.

Exclusion Criteria:

* Unwilling to take part in the study, or asked to be removed from the study at any time.
* History of alcohol intake > 20 g/day for 5 or more years
* Evidence autoimmune hepatitis, chronic hepatitis B or C virus, HIV, genetic hemochromatosis, alpha-1 antitrypsin deficiency, Wilson disease, or cirrhosis.
* Pregnancy.
* Currently taking known hepatotoxic medications.
* Failure to attend follow-up for a minimum of 1 year.
* Non-Saudi patients

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: NAFLD patients
Sampling Method: Non-Probability Sample
Enrollment: 35 (Estimated)
Dates: Start 2012-06; Primary Completion 2018-07 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Assessment of NAFLD histological changes after bariatric surgery (adjustable gastric banding, sleeve gastrectomy, gastric bypass, and duodenal switch). | Intra-operatively, 3 months and 1 year postoperatively.
  Histological evaluation is done by applying the NAFLD activity score (NAS). The stage of fibrosis will be determined by the five-point (stage 0 to 4) scale.

SECONDARY OUTCOMES:
Assessment of liver function after bariatric surgery. | Preoperatively, 3 months, 6 months, 1 year and annually for 5 year postoperatively.
  * Measure serum albumin, bilirubin, INR, anti-thrombin-III, ALT, GGT, AST, protein C and S levels.
  * Measure albumin synthesis using radiolabeled amino acids.
Assessment of NAFLD associated morbidities by detecting the systemic inflammatory changes after bariatric surgery. | preoperatively, 3 months, 6 months, 1 year and annually for 5 year postoperatively.
  - Study systemic inflammatory changes by measuring the serum levels of several inflammatory mediators: ESR, C-reactive protein, interleukins (IL-1, IL-4, IL-6, IL-8, IL-10, IL-16), adipokines (adiponectin, leptin, adipsin and Chemerin), MCP1, osteopontin, and growth factors (TNF-α, and VEGF).
Assessment of NAFLD associated morbidities by detecting the local inflammatory changes after bariatric surgery. | Baseline (tissues obtained intraoperatively).
  * Hepatic expression of α-SMA, collagen α1, TGF-β1, MCP-1, IL-6, IL-8, leptin and adiponectin receptors. PAI1, ACRP30, ADIPOQ.
  * Visceral adipose tissue to assess the expression of NOD-like receptor pyrin domain-containing-3 inflammasome (Nlrp3); are inflammatory markers that recognize certain signals that leads to caspase-1 activation and subsequent IL-1 and IL-18.
  * Subcutaneous adipose tissue to assess the expression of adiponectin, IL-6 and TNF-α.
Assessment of NAFLD associated morbidities by detecting the metabolic changes after bariatric surgery. | Preoperative, 3 months, 6 months, 1 year and annually for 5 years postoperatively.
  * Hormonal changes: serum levels of ghrelin, peptide YY, amylin, cholecystokinin, insulin, glucagon, epinephrine, and cortisol.
  * Non-hormonal changes: HbA1c, FFA, HDL, cholesterol, triglycerides, fasting glucose.
Assessment of NAFLD associated morbidities by detecting the endothelial changes after bariatric surgery. | Preoperative, 6 months, 1, 2 and 5 years postoperatively.
  * Doppler Ultrasound (Duplex) for the carotid arteries.
  * Measuring the levels of progenitor cells.
Studying the genetic factors expressing for the inflammatory changes differences in responders. | Baseline (for liver, visceral and subcutaneous fat). Postoperatively (for liver only): 3 months, 1 year and 5 years after the surgery.
  * TMA construction using the formalin stored liver, visceral fat and abdominal wall muscle.
  * Detecting mRNA expression from frozen tissue (liver, visceral fat and abdominal wall muscle) with respect of inflammation, insulin action, lipid metabolism, liver regression and apoptosis.
  * Deep gene sequencing for subgroup of patients with variables clinical responses or with genetic differences determined form the above testing.
Long-term follow-up to examine the correlation between the type of surgery and clinical outcomes associated with NAFLD (liver cirrhosis, incidence of cancer, and mortality). | 5 years
  Histological evaluation is done by applying the NAFLD activity score (NAS). The stage of fibrosis will be determined by the five-point (stage 0 to 4) scale.
Testing the efficacy of the non-invasive images in the diagnosis of NAFLD. | Baseline (preoperatively), 1 year and 5 years postoperatively.
  * Magnetic Resonance Studies.
  * Fibroscan.
  * Ultrasound.

CONTACTS AND LOCATIONS:
Overall Officials: Dr.Mazen Hassanain, MBBS FRCSC PhD, Principal Investigator — King Khalid University Hospital,King Saud University,Riyadh,KSA.
Locations (1):
- King Khalid University Hospital, Riyadh, Saudi Arabia

REFERENCES:
- [Background] Beymer C, Kowdley KV, Larson A, Edmonson P, Dellinger EP, Flum DR. Prevalence and predictors of asymptomatic liver disease in patients undergoing gastric bypass surgery. Arch Surg. 2003 Nov;138(11):1240-4. doi: 10.1001/archsurg.138.11.1240. PMID 14609874
- [Background] Gholam PM, Kotler DP, Flancbaum LJ. Liver pathology in morbidly obese patients undergoing Roux-en-Y gastric bypass surgery. Obes Surg. 2002 Feb;12(1):49-51. doi: 10.1381/096089202321144577. PMID 11868297
- [Background] Oliveira CP, Faintuch J, Rascovski A, Furuya CK Jr, Bastos Mdo S, Matsuda M, Della Nina BI, Yahnosi K, Abdala DS, Vezozzo DC, Alves VA, Zilberstein B, Garrido AB Jr, Halpern A, Carrilho FJ, Gama-Rodrigues JJ. Lipid peroxidation in bariatric candidates with nonalcoholic fatty liver disease (NAFLD) -- preliminary findings. Obes Surg. 2005 Apr;15(4):502-5. doi: 10.1381/0960892053723493. PMID 15946429
- [Background] Frantzides CT, Carlson MA, Moore RE, Zografakis JG, Madan AK, Puumala S, Keshavarzian A. Effect of body mass index on nonalcoholic fatty liver disease in patients undergoing minimally invasive bariatric surgery. J Gastrointest Surg. 2004 Nov;8(7):849-55. doi: 10.1016/j.gassur.2004.07.001. PMID 15531238
- [Background] Dixon JB, Bhathal PS, O'Brien PE. Nonalcoholic fatty liver disease: predictors of nonalcoholic steatohepatitis and liver fibrosis in the severely obese. Gastroenterology. 2001 Jul;121(1):91-100. doi: 10.1053/gast.2001.25540. PMID 11438497
- [Background] Ruhl CE, Everhart JE. Determinants of the association of overweight with elevated serum alanine aminotransferase activity in the United States. Gastroenterology. 2003 Jan;124(1):71-9. doi: 10.1053/gast.2003.50004. PMID 12512031
- [Background] Spaulding L, Trainer T, Janiec D. Prevalence of non-alcoholic steatohepatitis in morbidly obese subjects undergoing gastric bypass. Obes Surg. 2003 Jun;13(3):347-9. doi: 10.1381/096089203765887633. PMID 12841891
- [Background] Moretto M, Kupski C, Mottin CC, Repetto G, Garcia Toneto M, Rizzolli J, Berleze D, de Souza Brito CL, Casagrande D, Colossi F. Hepatic steatosis in patients undergoing bariatric surgery and its relationship to body mass index and co-morbidities. Obes Surg. 2003 Aug;13(4):622-4. doi: 10.1381/096089203322190853. PMID 12940291
- [Background] Silverman EM, Sapala JA, Appelman HD. Regression of hepatic steatosis in morbidly obese persons after gastric bypass. Am J Clin Pathol. 1995 Jul;104(1):23-31. doi: 10.1093/ajcp/104.1.23. PMID 7611176
- [Background] Dixon JB, Bhathal PS, Hughes NR, O'Brien PE. Nonalcoholic fatty liver disease: Improvement in liver histological analysis with weight loss. Hepatology. 2004 Jun;39(6):1647-54. doi: 10.1002/hep.20251. PMID 15185306
- [Background] Blackburn GL, Mun EC. Effects of weight loss surgeries on liver disease. Semin Liver Dis. 2004 Nov;24(4):371-9. doi: 10.1055/s-2004-860866. PMID 15605305
- [Background] Grimm IS, Schindler W, Haluszka O. Steatohepatitis and fatal hepatic failure after biliopancreatic diversion. Am J Gastroenterol. 1992 Jun;87(6):775-9. PMID 1590319
- [Background] Vandanmagsar B, Youm YH, Ravussin A, Galgani JE, Stadler K, Mynatt RL, Ravussin E, Stephens JM, Dixit VD. The NLRP3 inflammasome instigates obesity-induced inflammation and insulin resistance. Nat Med. 2011 Feb;17(2):179-88. doi: 10.1038/nm.2279. Epub 2011 Jan 9. PMID 21217695
- [Background] DeFronzo RA, Tobin JD, Andres R. Glucose clamp technique: a method for quantifying insulin secretion and resistance. Am J Physiol. 1979 Sep;237(3):E214-23. doi: 10.1152/ajpendo.1979.237.3.E214. PMID 382871
- [Background] Hompesch M, Rave K. An analysis of how to measure glucose during glucose clamps: are glucose meters ready for research? J Diabetes Sci Technol. 2008 Sep;2(5):896-8. doi: 10.1177/193229680800200522. PMID 19885275
- [Background] Mathurin P, Gonzalez F, Kerdraon O, Leteurtre E, Arnalsteen L, Hollebecque A, Louvet A, Dharancy S, Cocq P, Jany T, Boitard J, Deltenre P, Romon M, Pattou F. The evolution of severe steatosis after bariatric surgery is related to insulin resistance. Gastroenterology. 2006 May;130(6):1617-24. doi: 10.1053/j.gastro.2006.02.024. PMID 16697725
- [Background] Mathurin P, Hollebecque A, Arnalsteen L, Buob D, Leteurtre E, Caiazzo R, Pigeyre M, Verkindt H, Dharancy S, Louvet A, Romon M, Pattou F. Prospective study of the long-term effects of bariatric surgery on liver injury in patients without advanced disease. Gastroenterology. 2009 Aug;137(2):532-40. doi: 10.1053/j.gastro.2009.04.052. Epub 2009 May 4. PMID 19409898
- [Background] Moschen AR, Molnar C, Geiger S, Graziadei I, Ebenbichler CF, Weiss H, Kaser S, Kaser A, Tilg H. Anti-inflammatory effects of excessive weight loss: potent suppression of adipose interleukin 6 and tumour necrosis factor alpha expression. Gut. 2010 Sep;59(9):1259-64. doi: 10.1136/gut.2010.214577. Epub 2010 Jul 21. PMID 20660075
- [Background] Phillips ML, Boase S, Wahlroos S, Dugar M, Kow L, Stahl J, Slavotinek JP, Valentine R, Toouli J, Thompson CH. Associates of change in liver fat content in the morbidly obese after laparoscopic gastric banding surgery. Diabetes Obes Metab. 2008 Aug;10(8):661-7. doi: 10.1111/j.1463-1326.2007.00793.x. Epub 2007 Oct 17. PMID 17941875